CLINICAL TRIAL: NCT02505997
Title: A Phase I Study to Evaluate the Effect of Repeated Oral Doses of Delafloxacin on the Pharmacokinetics of a Single Oral Dose of Midazolam in Healthy Subjects
Brief Title: Study to Evaluate the Effect of Delafloxacin on the Pharmacokinetics of Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ML-3341-118
Record Dates: First submitted 2015-06-23; First posted 2015-07-22 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: VA Drug Interactions
MeSH Terms: interventions — Midazolam; delafloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Midazolam/Delafloxacin (Experimental): Each subject will receive a single 5 mg oral dose of midazolam syrup on Day 1, oral 450 mg delafloxacin tablets twice daily (Q12h) for Days 3 to 8, and co-administered a single 5 mg oral dose of midazolam syrup in the AM on Day 8.
  Interventions: Drug: Midazolam; Drug: Delafloxacin

INTERVENTIONS:
Drug: Midazolam — Single 5 mg oral dose of midazolam syrup given in the AM on Day 1 and Day 8.
Drug: Delafloxacin — Oral 450 mg delafloxacin tablets given twice daily (Q12h) on Days 3 to 8

SUMMARY:
The purpose of this study is to evaluate the effect of repeated doses of oral delafloxacin on the pharmacokinetic (PK) profile of a single oral dose of midazolam.

DETAILED DESCRIPTION:
This study will evaluate the effect of repeated doses of oral delafloxacin on the PK profile of a single oral dose of midazolam. The study will also evaluate the pharmacokinetics, safety, and tolerability of repeated oral doses of delafloxacin in healthy male and female subjects and to obtain a steady state PK profile for oral delafloxacin.

ELIGIBILITY:
Inclusion Criteria:

* No clinically important abnormal physical findings.
* No clinically significant laboratory abnormalities.
* Normal (or abnormal but not clinically significant) ECG measurements.
* Body mass index between 18.0 and 32.0 kg/m2.
* Normal (or abnormal but not clinically significant) blood pressure and pulse rate measurements. methylxanthine-containing beverages or food
* Non-smoker

Exclusion Criteria:

* Received any investigational drug within 8 weeks before administration of the first dose of the study drug
* Female who is pregnant, has a positive pregnancy test, or is breastfeeding.
* Positive test result for amphetamines, barbiturates, benzodiazepines, cocaine metabolites, opiates, cannabinoids, methylenedioxymethamphetamine, cotinine, or alcohol in urine at Screening or Day -1.
* Positive screening test for hepatitis B surface antigen, hepatitis C, and/or human immunodeficiency virus antibodies.
* Any surgical or medical condition that, in the judgment of the investigator, might interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Used any medication (prescription or over-the-counter, including health supplements and herbal remedies, with the exception of acetaminophen, as defined in exclusion number 8) within 2 weeks (4 weeks for drugs or substances known to inhibit or induce CYP enzymes and/or P-gp including St. John's wort [Hypericum perforatum]) or 5 half-lives (whichever is longer) before the first dose of study drug.
* Used an oral or IV antibiotic within 4 weeks of administration of the first dose of the study drug.
* Routinely or chronically used more than 2 g of acetaminophen daily.
* Performed strenuous activity, sunbathing, and/or contact sports within 96 hours (4 days) before entry into the clinical study site on Day -1, and for the duration of the study.
* Donated or lost greater than 400 mL of blood in the 30 days before administration of the first dose of the study drug.
* History of clinically significant GI disease, or gastroenteritis (vomiting or diarrhea) or any history of GI bleeding (excluding bleeding from hemorrhoids)
* History of any significant drug allergy
* History of any drug or alcohol abuse in the past 2 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Midazolam and 1-hydroxymidazolam Plasma PK: AUC0-t | Days 1 and 8
Midazolam and 1-hydroxymidazolam Plasma PK: AUC0-inf | Days 1 and 8
Midazolam and 1-hydroxymidazolam Plasma PK: Cmax | Days 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Sue Cammarata, MD, Study Director — Melinta Therapeutics, Inc.
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- [Derived] Paulson SK, Wood-Horrall RN, Hoover R, Quintas M, Lawrence LE, Cammarata SK. The Pharmacokinetics of the CYP3A Substrate Midazolam After Steady-state Dosing of Delafloxacin. Clin Ther. 2017 Jun;39(6):1182-1190. doi: 10.1016/j.clinthera.2017.04.009. Epub 2017 May 9. PMID 28495029